CLINICAL TRIAL: NCT03903458
Title: Open Label, Non-randomized, Phase IB Study to Characterize Safety, Tolerability and Recommended Dose of Tinostamustine and Nivolumab in Patients With Refractory, Locally Advanced or Metastatic MelAnoma
Brief Title: Tinostamustine and Nivolumab in Advanced Melanoma
Acronym: ENIgMA
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Markus Joerger (Other)
Responsible Party: Sponsor-Investigator, Markus Joerger, Chair Clinical Research Unit, Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTU 17.022
Record Dates: First submitted 2019-03-13; First posted 2019-04-04 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Malignant Melanoma
Keywords: systemic anticancer treatment; immunotherapy; epigenetic treatment
MeSH Terms: conditions — Melanoma | interventions — tinostamustine; Nivolumab

STUDY DESIGN:
Intervention Model Description: this is an open label, non-randomized, Phase IB clinical trial studying a new anticancer drug combination
Masking Description: open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tinostamustine and Nivolumab (Experimental): Experimental drug combination arm
  Interventions: Drug: Tinostamustine

INTERVENTIONS:
Drug: Tinostamustine — First-in-human administration of the combination of Tinostamustine and Nivolumab.
  Other Names: Nivolumab

SUMMARY:
This trial is a first-in-human drug combination with the first-in-class alkylating histone deacetylase inhibition (HDACi) fusion molecule Tinostamustine (EDO-S101) and the anti-PD-1 monoclonal antibody Nivolumab in patients with refractory, locally advanced or metastatic melanoma.

DETAILED DESCRIPTION:
Despite improvement of systemic treatment in patients with advanced melanoma, there is still unmet medical need in this group of patients. Tinostamustine is a medication without marketing authorization, while Nivolumab is approved for several tumor entities. The primary objective of this trial is to assesses the safety, tolerability and recommended dose of Tinostamustine in combination with Nivolumab in patients with advanced melanoma.Secondary objectives of this trial in patients with advanced solid tumors are to assess the preliminary efficacy of Tinostamustine when given in combination with Nivolumab and to characterize potential predictive biomarkers of the combination treatment of Tinostamustine and Nivolumab. The trial includeds patients with either histologically or cytologically confirmed inoperable stage III or metastatic stage IV melanoma with an indication for the regular systemic treatment with Nivolumab and a maximum of 1 prior systemic palliative line of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Patients with either histologically or cytologically confirmed inoperable stage III or metastatic stage IV melanoma
* Indication for the regular systemic treatment with the anti-PD-1 monoclonal antibody Nivolumab monotherapy
* Patient received a maximum of 1 prior systemic palliative line of treatment
* ECOG ≤2
* Patients with brain metastases must have undergone definitive treatment (surgery or radiotherapy) at least 2 weeks prior to starting study drug and be documented as having stable disease by imaging
* Adequate bone marrow, renal and hepatic function
* Adequate contraception

Exclusion Criteria:

* Prior treatment with a PD-(L)1 targeted monoclonal antibody
* Patients who have received systemic treatments or radiotherapy within 2 weeks prior to starting study drug
* Concomittant treatment with systemic steroids at a daily dose equivalent to ≥10mg of prednisone, or concomittant treatment with immunosuppressive drugs such as methotrexate
* Patients with a prior malignancy are excluded (except non-melanoma skin cancers, and in situ cancers such as the following: bladder, colon,cervical/dysplasia, melanoma, or breast). Patients with other second malignancies diagnosed more than 2 years ago who have received therapy with curative intent with no evidence of disease during the interval who are considered by the Investigator to present a low risk for recurrence will be eligible.
* NYHA stage III/IV congestive heart failure and/or arrhythmia not adequately controlled
* QTc interval (Fridericia's formula) > 450msec
* Patients who are on treatment with drugs known to prolong the QT/QTc interval (Credible Meds list:

Known risk of TdP. https://www.crediblemeds.org).

* Pregnant and breast feeding patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2019-03-07 (Actual); Primary Completion 2021-12-15 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
Safety and dose-limiting toxicity | at 6 weeks
  Dose limiting toxicity defined as any of the following AEs (according to CTCAE v 4.03) occurring during the first 42 days of study treatment for each study patient of the safety part of the trial, and regarded to be related (possibly, probably or definitely) to Tinostamustine:
  * CTC °4 neutropenia during ≥ 5 days
  * Febrile neutropenia
  * CTC °4 thrombocytopenia or CTC° 3 thrombocytopenia with bleeding
  * Any other ≥ CTC °4 hematological AE
  * ≥ CTC °3 AST or ALT elevations for >7 days, or CTC °4 AST/ALT elevations for any duration
  * ≥ CTC °3 nausea, vomiting or diarrhea despite appropriate pre-medication
  * Any other ≥ CTC °3 non-hematological study-treatment-related AE, excluding alopecia
  * ≥ CTC °3 uveitis, pneumonitis, bronchospasm, neurological toxicity, hypersensi-tivity reactions or infusion reactions that result in discontinuation of study treat-ment
  * Any study treatment-related AE that results in a delay of the administration of Tinostamustine of at least 4 weeks

SECONDARY OUTCOMES:
Overall safety profile of the tinostamustine/nivolumab drug combination | during a maximum 2 years of study treatment plus 100 days thereafter (3 years)
  All adverse events (AE) including laboratory safety parameters according to CTCAE v.4.03
Radiological response | every 8 weeks until progressive disease or end of study (5 years)
  Objective tumor response according to RECIST 1.1 and iRECIST
Progression-free survival | through study completion (5 years)
  Progression-free survival (PFS, iPFS), defined as the time between registration to the study and the time of disease progression according to RECIST v.1.1 and iRECIST or death of the patient, whatever occurs first
Overall survival | through study completion (5 years)
  Overall survival (OS) from registration of study participation

CONTACTS AND LOCATIONS:
Overall Officials: Markus Joerger, Prof., Study Chair — Cantonal Hospital of St. Gallen
Locations (2):
- Switzerland (2):
  - Kantonsspital Graubünden, Chur
  - Cantonal Hospital St.Gallen, Sankt Gallen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials Unit St. Gallen, Switzerland — https://www.kssg.ch/mfz/clinical-trials-unit-ctu